CLINICAL TRIAL: NCT04871932
Title: Evolution of Immune System in Healthy Adults After Vaccination of New Coronavirus (COVID-2019) Inactivated Vaccine Based on Single Cell Multi-Omics Technologies
Brief Title: COVID-2019 Vaccine Immune Response Base on Single Cell Multi-Omics
Status: Recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Jun Pu, Director of Cardiovascular Medicine, RenJi Hospital
Other Study IDs: COVID-2019-VIR-SCMO study
Record Dates: First submitted 2021-04-30; First posted 2021-05-04 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Immune System and Related Disorders
Keywords: Cohort study; Immune System; PBMC; China

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral venous blood samples from each donor were obtained to get the peripheral blood mononuclear cells (PBMCs)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Recently unvaccinated group (Female): This study intends to collect peripheral blood from healthy adults aged 18 to 50 years. Gender and vaccination may be independent potential factors that affect the changes in peripheral blood immune cells. This study collects basic clinical information from volunteers, and classifies the population based on gender and whether they have been vaccinated recently (including influenza vaccine, human papillomavirus [HPV] vaccine, and severe acute respiratory syndrome [SARS]-CoV-2 vaccines and others), aiming at systematically classify the peripheral blood mononuclear cells of healthy adults under different conditions and search for molecular markers related to different cell types. This group is Recently unvaccinated group (Female)．
- Recently unvaccinated group (Male): This study intends to collect peripheral blood from healthy adults aged 18 to 50 years. Gender and vaccination may be independent potential factors that affect the changes in peripheral blood immune cells. This study collects basic clinical information from volunteers, and classifies the population based on gender and whether they have been vaccinated recently (including influenza vaccine, HPV vaccine, and SARS-CoV-2 vaccines and others), aiming at systematically classify the peripheral blood mononuclear cells of healthy adults under different conditions and search for molecular markers related to different cell types. This group is Recently unvaccinated group (Male)．
- Recently vaccinated group (Female): This study intends to collect peripheral blood from healthy adults aged 18 to 50 years. Gender and vaccination may be independent potential factors that affect the changes in peripheral blood immune cells. This study collects basic clinical information from volunteers, and classifies the population based on gender and whether they have been vaccinated recently (including influenza vaccine, HPV vaccine, and SARS-CoV-2 vaccines and others), aiming at systematically classify the peripheral blood mononuclear cells of healthy adults under different conditions and search for molecular markers related to different cell types. This group is Recently vaccinated group (Female)．
  Interventions: Biological: Recently Vaccination
- Recently vaccinated group (Male): This study intends to collect peripheral blood from healthy adults aged 18 to 50 years. Gender and vaccination may be independent potential factors that affect the changes in peripheral blood immune cells. This study collects basic clinical information from volunteers, and classifies the population based on gender and whether they have been vaccinated recently (including influenza vaccine, HPV vaccine, and SARS-CoV-2 vaccines and others), aiming at systematically classify the peripheral blood mononuclear cells of healthy adults under different conditions and search for molecular markers related to different cell types. This group is Recently vaccinated group (Male)．
  Interventions: Biological: Recently Vaccination

INTERVENTIONS:
Biological: Recently Vaccination
  Groups: Recently vaccinated group (Female); Recently vaccinated group (Male)

SUMMARY:
In recent years, single-cell high-throughput sequencing technology has developed rapidly and is widely used in research related to the immune system, breaking traditional cognition and gaining a new understanding of immune cell classification. In particular, the emerging single cell RNA sequencing (scRNA-seq) provides new ideas for the study of cell heterogeneity in multicellular organisms. Analyzing the changes in the expression profile of the cell transcriptome at the single-cell level can clearly show the changes in the trajectory of individual cells, reveal new cell types, and discover the potential functions of immune cells. Therefore, this study intends to recruit healthy adults and use multi-omics techniques such as single-cell sequencing to systematically classify the peripheral blood mononuclear cells of healthy adults to provide a basis for further disease-related research.

DETAILED DESCRIPTION:
As an important part of the human body, the immune system is closely related to the occurrence of diseases. Based on the traditional classification methodology, it is mainly divided into two branches: innate immunity and adaptive immunity. Innate immune cells mainly include monocytes (Mono), natural killer (NK) cells and dendritic cells (DC). The adaptive immune cells mainly include B lymphocytes (B) and T lymphocytes (T). Peripheral blood mononuclear cells (PBMCs) mainly include T cells, B cells, NK cells, Mono cells and DC cells.

The proportion of these cell populations varies among individuals. Usually in PBMC, T lymphocytes account for 45-70%, B cells account for 5-15%, NK cells account for 5-20%, Mono cells account for 10-30%, and DC cells account for 1-2%. Among them, B cells can be divided into transitional, naive, memory subgroups and plasma cells. While, T cells are mainly composed of cluster of differentiation 4+ (CD4+) T cells and cluster of differentiation 8+ (CD8+) T cells with the ratio about 2:1. What's more, CD4+ T cells and CD8+ T cells can be further divided into naive cells, central memory cells in contact with antigen, effector memory cells and effector cells. Mono cells can be divided into classic monocytes and non-classical cluster of differentiation 16+ (CD16+) pro-inflammatory monocytes. DC cells include plasmacytic dendritic cells (pDC) and myeloid dendritic cells (mDC).

In recent years, scRNA-seq has developed rapidly and is widely used in research related to the immune system, breaking traditional cognition and gaining a new understanding of immune cell classification. In particular, the emerging scRNA-seq provides new ideas for the study of cell heterogeneity in multicellular organisms. Analyzing the changes in the expression profile of the cell transcriptome at the single-cell level can clearly show the changes in the trajectory of individual cells, reveal new cell types, and discover the potential functions of immune cells.

Adults have a relatively stable immune system, with little interference from the external environment. Therefore, this study intends to recruit healthy adults and use multi-omics techniques such as scRNA-seq to systematically classify the PBMCs of healthy adults to provide a basis for further disease-related research.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 50 years; 2. No history of major diseases, no history of bacterial or viral infection in the past 3 months; 3. No recent history of surgery or trauma; 4 No history of smoking or alcoholism; 5. No immune system disease.

Exclusion Criteria:

1. Infectious diseases; 2. Tumor diseases; 3. Hematological diseases; 4. History of hypertension and diabetes; 5 Autoimmune diseases; 6 History of liver and kidney insufficiency; 7. History of previous cardiovascular diseases; 8. Pregnancy Or breast-feeding; 9. Past and current use of immunosuppressive drugs

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adults with Han nationality
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2026-11-03 (Estimated); Study Completion 2026-12-03 (Estimated)

PRIMARY OUTCOMES:
Changes in classification of human peripheral blood mononuclear cells | up to five years
  The primary endpoint will be the changes in classification of human peripheral blood mononuclear cells at single cell resolution.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Pu, MD,PhD, Principal Investigator — Cardiology, Ren Ji Hospital Shanghai, China
Locations (1):
- Cardiology, Ren Ji Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tong R, Luo L, Zhao Y, Sun M, Li R, Zhong J, Chen Y, Hu L, Li Z, Shi J, Lyu Y, Hu L, Guo X, Liu Q, Shuang T, Zhang C, Yuan A, Sun L, Zhang Z, Qian K, Chen L, Lin W, Chen AF, Wang F, Pu J. Characterizing the cellular and molecular variabilities of peripheral immune cells in healthy recipients of BBIBP-CorV inactivated SARS-CoV-2 vaccine by single-cell RNA sequencing. Emerg Microbes Infect. 2023 Dec;12(1):e2187245. doi: 10.1080/22221751.2023.2187245. PMID 36987861